CLINICAL TRIAL: NCT00095732
Title: A Phase 2, Randomized, Double Blind, Parallel Dose Ranging Study of Oral TheraCLEC™ - Total in Cystic Fibrosis Subjects With Exocrine Pancreatic Insufficiency
Brief Title: Oral TheraCLEC™ - Total in Cystic Fibrosis Subjects With Exocrine Pancreatic Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14269; I5L-MC-TCAA (Other: Eli Lilly and Company); TC-2A (Other: Altus/Alnara)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis; Pancreatic Insufficiency
Keywords: Pancreatic Insufficiency; Cystic Fibrosis; Enzymes
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — liprotamase lipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Liprotamase Dose (Experimental): Liprotamase in a fixed combination of lipase (5,000 units), protease (5,000 units) and amylase (750 units) administered orally (one Size 5 capsule of liprotamase and five Size 2 capsules of placebo) with each of three meals and two snacks daily for 28 days
  Interventions: Drug: Liprotamase; Drug: Placebo
- Mid Liprotamase Dose (Experimental): Liprotamase in a fixed combination of lipase (25,000 units), protease (25,000 units) and amylase (3,750 units) administered orally (one Size 5 capsule of liprotamase, one Size 2 capsule of liprotamase, and four Size 2 capsules of placebo) with each of three meals and two snacks daily for 28 days
  Interventions: Drug: Liprotamase; Drug: Placebo
- High Liprotamase Dose (Experimental): Liprotamase in a fixed combination of lipase (100,000 units), protease (100,000 units) and amylase (15,000 units) administered orally (one Size 5 capsule of placebo and five Size 2 capsules of liprotamase) with each of three meals and two snacks daily for 28 days
  Interventions: Drug: Liprotamase; Drug: Placebo

INTERVENTIONS:
Drug: Liprotamase — Administered orally as either Size 2 capsules (20,000 Units lipase; 20,000 Units protease; and 3,000 Units amylase) or Size 5 capsules (5,000 Units lipase; 5,000 Units protease; and 750 Units amylase)
  Other Names: ALTU-135; LY3031642; TheraCLEC - Total
Drug: Placebo — Administered orally in either Size 2 or Size 5 capsules

SUMMARY:
The purpose of this study is to determine the most effective dose of a new enzyme therapy on oral nutrient absorption in cystic fibrosis (CF) subjects with exocrine pancreatic insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic insufficiency (PI) documented by fecal elastase <100 mcg/gram measured at screening
* Diagnosis of CF based upon the following criteria:

  * two clinical features consistent with CF AND
  * either genotype with two identifiable mutations consistent with CF OR
  * sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis
* Forced Expiratory Volume Over One Second (FEV1) ≥30% predicted
* Clinically stable with no evidence of acute upper or lower respiratory tract infection

Exclusion Criteria:

* Pregnancy, breastfeeding or of childbearing potential and/or not willing to use accepted methods of birth control during enrollment in the study
* History of fibrosing colonopathy
* History of liver transplant or lung transplant
* Unable to discontinue enteral tube feedings during the study
* Subject weight <40 kg
* Known hypersensitivity to food additives
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to screening
* Unable to discontinue the use of pancreatic enzymes for a 72-hour period or any other condition that the investigator believes would interfere with the intent of this study or would make study participation not in the best interest of the subject

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2004-06; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline up to 19 days in Coefficient of fat absorption (CFA) | Baseline, up to 19 days

SECONDARY OUTCOMES:
Change from baseline up to 19 day in Coefficient of nitrogen absorption (CNA) | Baseline, up to 19 days
Change from baseline up to 19 days in stool weight | Baseline, up to 19 days
Change from baseline to 29 day endpoint in Cystic Fibrosis Questionnaire (CFQ) scale scores | Baseline, 29 days
Change from baseline up to 19 days in number of Stools | Baseline, up to 19 days
Change from baseline to 28 days in maximum change in glucose response | Baseline through 28 days

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morgantown, West Virginia